CLINICAL TRIAL: NCT00622479
Title: Mechanistic Evaluations on Sorafenib Induced Hypophosphatemia in Patients With Advanced Renal Cell Carcinoma
Brief Title: Mechanistic Evaluation on Sorafenib Induced Hypophosphatemia.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12345
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: Sorafenib; Hypophosphatemia; Left ventricular ejection fraction (LVEF); Beta-type Natriuretic Peptide (BNP)
MeSH Terms: conditions — Carcinoma, Renal Cell; Hypophosphatemia | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib will be administered at 400mg BID for a 28 day cycle.

SUMMARY:
The purpose of this study is to:

1. To elucidate the mechanism involved in the sorafenib-induced hypophosphatemia and possible early effect of hypophosphatemia on bone mineral density
2. A secondary objective to assess the effect sorafenib treatment on evaluate left ventricular function (LVEF) and Beta-type natriuretic peptide in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Histologically or cytologically confirmed advanced RCC
* Evaluable disease with lesions measured by CT-scan or MRI according to modified Response Evaluation Criteria in Solid Tumors (RECIST)
* ECOG Performance Status of 0 or 1
* Adequate bone marrow, liver and renal functions as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin > 9.0 g/dL 1. Age greater Than 18 yrs old
  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Platelet count 100,000/mm3
  * Total bilirubin <= 1.5 times the upper limit of normal
  * ALT and AST <= 2.5 x upper limit of normal (<= 5 x upper limit of normal for patients with liver involvement of their cancer)
  * Amylase and lipase < 1.5 x the upper limit of normal
  * PT-INR/PTT 1.5 x ULN (Patients who are being prophylactically anti-coagulated with an agent such as coumadin or low molecular weight heparin or therapeutically anti-coagulated with LMWH will be allowed to participate provided that they meet these criteria; in addition, these patients must be monitored at appropriate intervals throughout study)
  * Serum creatinine < 2.0 x the upper limit of normal or creatinine clearance (CrCl) 45 mL/min (CrCl = Wt (kg) (140-age)/72 Cr level, female 0.85) for patients with creatinine levels above 2.0 x ULN
  * Phosphate 2.0 mg/dl
  * LVEF >/= 40%
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Negative results must be available prior to study treatment
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including the 30 day period after last study drug dosing. The investigator should advise the patient how to achieve adequate contraception
* Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Patients who meet the following criteria at the time of screening will be excluded:

  * History of cardiac disease: congestive heart failure >NYHA Class 2; hospitalization for CHF symptoms in the 6 months prior to study entry; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
  * Known history of HIV infection or chronic hepatitis B or C
  * Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
  * Active clinically serious infections (> Grade 2 CTCAE v3)
  * Known history or presence of metastatic brain or meningeal tumors (head CT or MRI at screening to confirm)
  * Patients with seizure disorder requiring medication (such as steroids or anti epileptics)
  * History of organ allograft
  * Patients undergoing renal dialysis
  * Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry
  * Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry. Mitomycin C or nitrosureas should not be given within 6 weeks of study entry. Anticancer therapy is defined as any agent or combination of agents with clinically proven anticancer activity administered by any route with the purpose of affecting the cancer, either directly or indirectly, including palliative and therapeutic endpoints
  * Radiotherapy to target lesions within 4 weeks of start of study drug
  * Major surgery within 4 weeks of start of study
  * Serious, non-healing wound, ulcer, or bone fracture
  * Investigational drug therapy within 4 weeks of study entry
  * Prior exposure to sorafenib
  * Pregnant or breast-feeding patients
  * Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
  * Known or suspected allergy to the investigational agent or any agent given in association with this trial
  * Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
  * Unable to swallow oral medications
  * Any malabsorption condition
  * Current treatment with bisphosphonates therapy or prior therapy with such agents within 12 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To evaluate a potential mechanism of hypophosphatemia related to sorafenib treatment based on measurement of phosphate regulating factors, peptides, and related laboratory variables | Occur when the last query is resolved

SECONDARY OUTCOMES:
To assess the effect of sorafenib treatment on left ventricular ejection fraction (LVEF) and B-type Natriuretic Peptide (BNP) in plasma | Occur when the last query is resolved

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (7):
  - Scottsdale, Arizona
  - Jacksonville, Florida
  - Maywood, Illinois
  - Detroit, Michigan
  - Rochester, Minnesota
  - Hackensack, New Jersey
  - Stony Brook, New York